CLINICAL TRIAL: NCT01564875
Title: Efficacy and Safety of Morning Intake of Simvast Controlled Release (CR) Tablet Versus Evening Intake of Zocor Tablet in Chronic Kidney Disease Stage(CKD)3, 4 and 5 Patients With Hyperlipidemia: A Randomized, Double-blind, Multicenter Phase 4 Trial (HM-SIM4)
Brief Title: Efficacy and Safety of Simvast Controlled Release (CR) and Zocor in Chronic Kidney Disease(CKD) Stage 3, 4 and 5 Patients With Hyperlipidemia
Acronym: HM-SIM4
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-SIM4
Record Dates: First submitted 2012-03-23; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Kidney Disease; Hyperlipidemia
Keywords: Simvast CR; Zocor
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperlipidemias | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvast CR (Experimental): * Simvast CR Tab 20mg, 1 tablet once daily to be administered between 6 and 9 a.m.
  * Placebo with the same appearance and formulation as that of Zocor Tab, 1 tablet once daily to be administered between 6 and 9 p.m.
  Interventions: Drug: Simvast CR
- Zocor (Active Comparator): * Placebo with the same appearance and formulation as that of Simvast CR Tab, 1 tablet once daily to be administered between 6 and 9 a.m.
  * Zocor Tab 20mg, 1 tablet once daily to be administered between 6 and 9 p.m.
  Interventions: Drug: Zocor

INTERVENTIONS:
Drug: Simvast CR — Simvast CR Tab 20mg, 1 tablet once daily to be administered between 6 and 9 a.m.
  Arms: Simvast CR
Drug: Zocor — Zocor Tab 20mg, 1 tablet once daily to be administered between 6 and 9 p.m.
  Arms: Zocor

SUMMARY:
Study design

* Multicenter, double-dummy, double-blinded, randomized, Phase 4 study
* Patients will be randomized to either a study group or a control group in a 1:1 ratio, and will be orally administered the assigned drugs

Study Objective

-The study is designed to demonstrate that efficacy and safety of morning dosing of Simvast Controlled Release (CR) Tab is not inferior to evening dosing of Zocor Tab in patients with stage 3,4,5 chronic kidney disease with hyperlipidemia

Primary objective

-to assess the percent change of LDL-C at Week 8 from baseline in Chronic Kidney Disease(CKD) stage 3,4,5 with hyperlipidemia subjects.

DETAILED DESCRIPTION:
The secondary objectives of the study are as follows:

* to assess the change and percent change of TC, HDL-C, TG from baseline.
* to assess the accomplishment rate of therapeutic goals based on the therapeutic guidance for hyperlipidemia of the Korean Society of Lipidology and Atherosclerosis.

ELIGIBILITY:
Inclusion criteria:

* Patient with age of 20 to 75 (inclusive)
* Patients with fasting serum lipid panels meeting the followings:

  * At Visit 1 screening 100mg/dL ≤ LDL-C < 220 mg/dL Triglyceride < 400mg/dL However, if the patient has been treated with antihyperlipidemics for 4 consecutive weeks or longer at the time of screening, it should be 100mg/ dL ≤ LDL-C < 160 mg/dL.
  * At Visit 2 screening 100mg/dL ≤ LDL-C < 220 mg/dL Triglyceride < 400mg/dL
* Patients with CKD stage 3 to 5.
* Subjects considered requiring medication by the principal investigator based on the therapeutic -guidance for hyperlipidemia of the Korean Society of Lipidology and Atherosclerosis.
* Patients who understand the study procedures and signed the informed consent form.

Exclusion criteria:

* Patients with a hypersensitivity to HMG-CoA reductase inhibitor or any of its ingredients.
* Patients who consume more than 14 units of alcohol a week, who are considered to have a history of drug overdose within 12 months of screening by the investigator, or who abuse other drugs.
* Patients with the following history:

  * Active gallbladder disease within 12 months of screening (patients who had cholecystectomy are eligible for the study).
  * Pancreatitis or liver disease (AST or ALT > 2 times the upper limit of the normal range at Visits 1 and 2).
  * Patients with uncontrolled diabetes mellitus (HbA1c ≥ 9.0 %).
  * Patients with hypotension (systolic blood pressure< 90mmHg or diastolic blood pressure<50mmHg).
  * Patients with uncontrolled hypertension: mean systolic blood pressure (SBP)> 160mmHg or mean diastolic blood pressure (DBP) > 100mmHg at Visit 2.
  * Patients with myocardial infarction or who had coronary artery bypass or angioplasty within 6 months before screening.
  * Patients who had stroke, transient ischemic attack (TIA), or deep vein thrombosis (DVT) within 6 months of screening.
  * Patients who had been treated for carotid artery disease, peripheral artery disease, or abdominal aortic aneurysm.
  * Patients with serious heart disease (patients with NYHA class (Attachment 4) III or IV congestive heart failure, unstable angina pectoris, or acute myocardial infarction).
  * Patients who were diagnosed with malignancy within 5 years or who have active tumors.
  * Patients with fibromyalgia, myopathy, rhadomyolysis, or sudden muscle pain, or patients who experienced adverse events during the previous treatment with statins.
  * Patients with mental illnesses considered by the investigator serious enough to adversely affect the patients' participation in the study.
  * Patients with uncontrolled primary hypothyroidism.
  * Patients with active peptic ulcer disease.
  * Patients with gastrointestinal conditions that may restrict drug absorptions, such as chronic diarrhea, inflammatory colic disease, partial ileal bypass, gastrorrhaphy, or gastric banding.
  * Screening CPK level > 3 times the upper limit of the normal range.
  * Patients on immunosuppressives after kidney transplantation.
  * Patients who need to be on immunosuppressives for other reasons.
* Patients who have participated in another clinical trial within the last 4 weeks of screening (except those who participated in clinical trials including observational studies that do not involve interventions such as medication).
* Pregnant women, lactating women, or women of childbearing potential who do not use appropriate contraceptives.
* Patients currently on dialysis.
* Other patients considered ineligible by the principal investigator and investigators.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Percent change of LDL-C | 8 weeks
  Percent change of LDL-C at Week 8 from baseline

SECONDARY OUTCOMES:
Change and percent change of TC, HDL-C, TG | 8 weeks
  Change and percent change of TC, HDL-C, TG from baseline.
Accomplishment rate of therapeutic goals | 8 weeks
  -Accomplishment rate of therapeutic goals based on the therapeutic guidance for hyperlipidemia of the Korean Society of Lipidology and Atherosclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-mi Park, Ph.D, Study Director — Hanmi Pharmaceutical Company Limited ( e-mail: kmpark@hanmi.co.kr )
Locations (7):
- South Korea (7):
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Eulji General Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702